CLINICAL TRIAL: NCT04501250
Title: A Double-blinded, Randomized, Comparative, Crossover Pharmacokinetics Study of Rinsulin® NPH, Suspension for Subcutaneous Administration, 100 IU/ml (GEROPHARM LLC, Russia) and Humulin® NPH, Suspension for Subcutaneous Administration, 100 IU/ml (Lilly France, France) Using Method of Euglycemic Hyperinsulinemic Clamp on Healthy Volunteers
Brief Title: Comparative Study of Rinsulin® NPH, Suspension for Subcutaneous Administration, 100 IU/ml (GEROPHARM LLC, Russia) and Humulin® NPH, Suspension for Subcutaneous Administration, 100 IU/ml (Lilly France, France) Using the Euglycemic Hyperinsulinemic Clamp Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RINCL-NPH
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Pharmacokinetics; Bioequivalence
Keywords: human recombinant insulin; euglycemic hyperinsulinemic clamp
MeSH Terms: interventions — Isophane Insulin, Human

STUDY DESIGN:
Intervention Model Description: Crossover Assignment two-way crossover
Who Masked: Participant, Investigator
Masking Description: A double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rinsulin® NPH (Experimental): Single subcutaneous administration of Insulin at a dose 0.4 IU / kg
  Interventions: Drug: Rinsulin NPH; Drug: Humulin NPH
- Humulin® NPH (Active Comparator): Single subcutaneous administration of Insulin at a dose 0.4 IU / kg
  Interventions: Drug: Rinsulin NPH; Drug: Humulin NPH

INTERVENTIONS:
Drug: Rinsulin NPH — subcutaneous injection at a dose of 0.4 IU/kg
Drug: Humulin NPH — subcutaneous injection at a dose of 0.4 IU/kg

SUMMARY:
Сomparative pharmacokinetic study of Rinsulin® NPH, suspension for subcutaneous administration, 100 IU/ml (GEROPHARM LLC, Russia) and Humulin® NPH, suspension for subcutaneous administration, 100 IU/ml (Lilly France, France) using the euglycemic hyperinsulinemic clamp.

DETAILED DESCRIPTION:
A double-blinded, randomized, comparative, crossover pharmacokinetics study of Rinsulin® NPH, suspension for subcutaneous administration, 100 IU/ml (GEROPHARM LLC, Russia) and Humulin® NPH, suspension for subcutaneous administration, 100 IU/ml (Lilly France, France) using method of euglycemic hyperinsulinemic clamp on healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Men of the Caucasian race with a verified diagnosis "healthy" according to the data of standard clinical, laboratory and instrumental examination methods.
* Age 18-50, inclusive.
* Body mass index 18.5 - 27 kg / m2.
* Volunteers who have sexual contact with fertile women should agree to use barrier methods of contraception while participating in the study (unless they have undergone surgical sterilization). Study Participants must also not become a sperm donor within the specified period.
* Consent to all restrictions imposed during the study.

Exclusion Criteria:

* Acute inflammatory diseases within 3 weeks from the moment of complete recovery to the stage of screening.
* Presence of episodes of hypoglycemia in the history of the volunteer
* Presence in the family history of the closest relatives cases of verified diagnosis of diabetes mellitus of any type.
* Deviations from the norm of basic vital indicators (heart rate, blood pressure, respiratory rate, body temperature) and ECG from normal values and laboratory values from reference values during screening.
* Fasting plasma glucose> 6.1 mmol / L at screening.
* HbA1C> 6% at the time of screening.
* Oral glucose tolerance test - blood glucose level ≥7.8 mmol / L (2 hours after glucose loading) during screening.
* Hard-to-reach veins of the upper extremities, vein thrombosis, history of thrombophlebitis or family history of close relatives, "compromised" veins due to frequent preceding venipuncture.
* Taking medications, phytopreparations, biologically active additives within 14 days before screening.
* Significant blood loss 3 months before screening due to, for example, but not limited to the following points: a. donor blood donation; b. extended surgery or trauma leading to significant blood loss.
* Incomplete recovery from surgery or surgery scheduled while the volunteer is participating in the study.
* Mental, physical and other reasons interferes with adequately assessing behavior and correctly fulfill the conditions of the research protocol (incl. a history of mental illness).
* Presence or history (three years before the the study drug) of narcotic, drug and / or substance abuse.
* Positive test for the content of narcotic drugs in urine during the screening period.
* Anamnestic information about alcoholism or taking more than 10 units. alcohol per week (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of dry wine or 50 ml of spirits).
* Positive test for alcohol in breath during screening.
* Nicotine addiction (regular use of tobacco less than 6 months before screening).
* Any chronic diseases, incl. but not limited to positive test results for hepatitis C or hepatitis B, HIV, syphilis at the time of screening.
* Burdened allergological history.
* presence of suspicion of an inflammatory disease of the urinary system based on the results of urinalysis during screening.
* Presence of oncological diseases within 5 years before the screening.
* History of organ transplantation (except of corneal transplant performed more than 3 months before the first injection of the study drug).
* Participation in a clinical trial of any drug or experimental medical device within 3 months prior to the first administration of the study drug.
* Any other condition that, in the reasonable opinion of the research physician, makes it difficult for the volunteer to participate in the study.
* History of hypersensitivity to heparin, insulin or any of the excipients of the investigational drugs.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Смах | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Test Drug Observed Maximum Plasma Concentration (Cmax)
AUC 0-12 | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 12 h
AUC GIR 0-12 | -2, -1.5, 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 12 h
AUC GIR 0-24 | -2, -1.5, 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 24 h
GIRmax | -2, -1.5, 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Maximum glucose infusion rate over the study period
tGIRmax | -2, -1.5, 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Time to reach maximum glucose infusion rate
tGIRlag | -2, -1.5, 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Time between the drug administration and the onset of action

SECONDARY OUTCOMES:
AUC 0-2 | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 2 h
AUC 0-6 | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 6 h
AUC 0-24 | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 24 h
AUC 0-∞ | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to ∞
Tmax | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Time to reach test drug Maximum Plasma Concentration
T1/2 | - 1 , -0.5 , 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24 hours
  Half-life of a drug tested

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Mr Noskov, AP of medicine, Principal Investigator — Yaroslavl City Clinical Hospital No. 3
Locations (1):
- Yarosslavl Clinical Hospital #3, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No